CLINICAL TRIAL: NCT00504127
Title: A Phase 3, 53 Weeks Study on Analgesic Efficacy and Safety of Naproxcinod (HCT 3012): 26-Week, Randomized, Parallel-Group, Double-Blind, Placebo (13 Weeks)- and Naproxen (26 Weeks)-Controlled, Multicenter Study of Naproxcinod (375 mg Bid and 750 mg Bid) With a 26-Week Naproxen-Controlled Safety Follow-up in Subjects With Osteoarthritis of the Knee, and a 1-week Post-treatment Safety Follow-up
Brief Title: Efficacy and Safety Study of Naproxcinod in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: Dr Brigitte Duquesroix, senior Director of Clinical Research, nicox
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCT 3012-X-302
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Degenerative
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — naproxen-n-butyl nitrate; BID protein, human; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- naproxcinod 375 mg bid (Experimental)
  Interventions: Drug: Naproxcinod 375 mg bid
- naproxcinod 750 mg bid (Experimental)
  Interventions: Drug: Naproxcinod 750 mg bid
- naproxen 500 mg bid (Active Comparator)
  Interventions: Drug: Naproxen 500 mg bid
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Naproxcinod 375 mg bid — Naproxcinod 375 mg bid
  Arms: naproxcinod 375 mg bid
Drug: Naproxcinod 750 mg bid — Naproxcinod 750 mg bid
  Arms: naproxcinod 750 mg bid
Drug: Naproxen 500 mg bid — Naproxen 500 mg bid
  Arms: naproxen 500 mg bid
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
To study of efficacy and safety of Naproxcinod vs. Naproxen and Placebo in the indication of signs and symptoms of osteoarthritis

DETAILED DESCRIPTION:
This is a 53 week study consisting in a 26 week randomized, double-blind, parallel group, multicenter study comparing efficacy and safety of Naproxcinod, Placebo and Naproxen. The first 26 weeks will be followed by a naproxen-controlled treatment period up to 52 weeks and a 1-week post-treatment safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men and Woman (40 or older) with a diagnosis of primary OA of the knee.
* Must be a current chronic user of NSAIDS or acetaminophen
* Must discontinue all analgesic therapy at Screening

Exclusion Criteria:

* Uncontrolled Hypertension or Diabetes
* Hepatic or Renal Impairment
* Current or expected use of anti-coagulant
* Clinical relevant abnormal ECG
* A history of alcohol or drug abuse
* Candidates for imminent joint replacement
* Participation within 30 days prior to screening in another investigational study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To show that both doses of Naproxcinod (375 mg twice daily [bid] and 750 mg bid) were superior to placebo in relieving osteoarthritis (OA) signs and symptoms in subjects with OA of the knee at Week 13. | 13 weeks

SECONDARY OUTCOMES:
To assess the efficacy of naproxcinod compared to naproxen 500 mg bid in relieving OA signs and symptoms in subjects with OA of the knee | 52 weeks
To evaluate the effect on blood pressure (BP) of both doses of naproxcinod, placebo, and naproxen 500 mg bid, as measured by the office BP monitoring in a population of OA subjects | 52 weeks
To obtain information regarding the pharmacokinetics/exposure of both doses of naproxcinod through a population pharmacokinetics (PK) approach | 52 weeks
To assess if there were any radiological changes at Week 52 in naproxcinod compared with naproxen subjects (target joint radiographs were taken at Screening and after 52 weeks of treatment, or if early termination occurred after Week 26) | 52 weeks
To compare the general safety and tolerability of both doses of naproxcinod versus naproxen 500 mg bid up to 52 weeks and with one Week post treatment follow up (Week 53) | 53 weeks

CONTACTS AND LOCATIONS:
Locations (73):
- United States (73):
  - Chandler, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Encino, California
  - Foothill Ranch, California
  - Orange, California
  - Rancho Mirage, California
  - Riverside, California
  - Denver, Colorado
  - Waterbury, Connecticut
  - Boca Raton, Florida
  - Brooksville, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Ocala, Florida
  - Pinellas Park, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Rockford, Illinois
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Erlanger, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Owings Mills, Maryland
  - Wellesley Hills, Massachusetts
  - Ann Arbor, Michigan
  - Brooklyn Center, Minnesota
  - Edina, Minnesota
  - Florissant, Missouri
  - St Louis, Missouri
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Columbus, Ohio
  - Marion, Ohio
  - Clinton, Oklahoma
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Anderson, South Carolina
  - Clinton, South Carolina
  - Goose Creek, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Cordova, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Garland, Texas
  - Houston, Texas
  - Nederland, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Lakewood, Washington